CLINICAL TRIAL: NCT05024227
Title: Discussion on the Effect of Nursing Education Intervention on Women's Health Literacy of Plasticizers
Brief Title: The Effect of Nursing Education Intervention on Women's Health Literacy of Plasticizers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, PhD, RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHGH-IRB:(864)110-10
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Endocrine Disrupting Chemicals; Health Literacy
Keywords: nursing education intervention; health literacy; plasticizers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: nursing education interventions (Experimental): nursing education interventions (including e-health platform assistance)
  Interventions: Behavioral: Experimental: nursing education interventions (including e-health platform assistance)
- No Intervention: Routine care (No Intervention): Only the original form of nursing education leaflets are given

INTERVENTIONS:
Behavioral: Experimental: nursing education interventions (including e-health platform assistance) — Nursing education intervention: Researchers use teaching, consultation and other methods to give individual cases planned learning to meet individual needs, providing 1. What is an environmental hormone-plasticizer; 2. Common types of environmental hormones (such as plasticizers) and Uses 3. Environmental hormones-sources of plasticizers 4. Environmental hormones-plasticizers harm to the human body 5. How to avoid the common environmental hormones-plasticizers and other related health education in life, and use the electronic platform to assist nursing education conduct.
  Arms: Experimental: nursing education interventions

SUMMARY:
Environmental hormone (environmental hormone), also known as "endocrine disrupting chemicals" (EDCS), is a pollutant that affects the endocrine system and causes diseases and dysfunction throughout the life cycle. Many daily products are ubiquitous, and the most common are phthalates (plasticizers); in recent years, many scientific research reports have determined the adverse health effects of phthalates, including: Infertility (Den Hond et al. al., 2015), testicular hypoplasia (Fisher, 2004), obesity (Dirtu et al., 2013), diabetes (Fénichel & Chevalier, 2017), hyperglycemia (Williams et al., 2016), asthma (Wang et al., 2016) al., 2015), endometriosis and high abortion rate (Roy et al., 2015), polycystic ovary syndrome (Vagi et al., 2014), prostate cancer (Chuang et al., 2020), and Breast cancer (Chen et al., 2020; Fu et al., 2017; Holmes et al., 2014; López-Carrillo et al., 2010), etc. In 2011, the Taiwan Food and Drug Administration detected di（2-ethylhexyl）phthalate (DEHP) and dibutyl phthalate (DBP) in foods, food supplements, and beverages, and determined that the Taiwanese population has a high content of phthalates (Yang et al., 2013). It pointed out that exposure to plasticizers in the uterus will have lifelong effects and even endanger the health of the next generation, indicating that there is a significant positive correlation between the concentration of metabolites in the urine of pregnant women and the urine of their children (Lin et al., 2011; Wu et al., 2013), even related to children's autism (Carter & Blizard, 2016; Rossignol et al., 2014).

However, so far there is still a lack of research on environmental hormone-plasticizers to improve health literacy or develop interventional research. Therefore, this study hopes to track the health literacy of their plasticizers and provide nursing education interventions (including e-health platform assistance) for women. Randomized controlled trials (English: randomized controlled trial, RCT) will be used to test nursing education interventions using a double-blind trial system. (Including e-health platform assistance) Effectiveness, in order to provide simple and fast self-health monitoring and management for the people, and it is expected that the case can early prevent the occurrence of related diseases and ensure the safety of the living environment.

DETAILED DESCRIPTION:
Environmental hormone (environmental hormone), also known as "endocrine disrupting chemicals" (EDCS), is a pollutant that affects the endocrine system and causes diseases and dysfunction throughout the life cycle. Many daily products are ubiquitous, and the most common are phthalates (plasticizers); in recent years, many scientific research reports have determined the adverse health effects of phthalates, including: Infertility (Den Hond et al. al., 2015), testicular hypoplasia (Fisher, 2004), obesity (Dirtu et al., 2013), diabetes (Fénichel & Chevalier, 2017), hyperglycemia (Williams et al., 2016), asthma (Wang et al., 2016) al., 2015), endometriosis and high abortion rate (Roy et al., 2015), polycystic ovary syndrome (Vagi et al., 2014), prostate cancer (Chuang et al., 2020), and Breast cancer (Chen et al., 2020; Fu et al., 2017; Holmes et al., 2014; López-Carrillo et al., 2010), etc. In 2011, the Taiwan Food and Drug Administration detected DEHP and DBP in foods, food supplements, and beverages, and determined that the Taiwanese population has a high content of phthalates (Yang et al., 2013). It pointed out that exposure to plasticizers in the uterus will have lifelong effects and even endanger the health of the next generation, indicating that there is a significant positive correlation between the concentration of metabolites in the urine of pregnant women and the urine of their children (Lin et al., 2011; Wu et al., 2013), even related to children's autism (Carter & Blizard, 2016; Rossignol et al., 2014).

Health literacy is an important factor in determining public and personal health, and is regarded as the core of patient-centered care. Relevant studies have indicated that a lack of health literacy has the following results: higher mortality, poor self-management skills, lower satisfaction with medical and disease communication, poor awareness of diseases, higher hospitalization and emergency medical use rates, easier incorrect medication, low utilization of preventive health care services (such as screening), high prevalence of chronic diseases (such as cardiovascular disease, diabetes, and obesity, etc.), and high health care costs (Berkman, Sheridan, Donahue, Halpern, & Crotty, 2011; Berkman, Sheridan, Donahue, Halpern, Viera, et al., 2011; DeWalt et al., 2004). However, so far there is still a lack of research on environmental hormone-plasticizers to improve health literacy or develop interventional research. Therefore, this study hopes to track the health literacy of their plasticizers and provide nursing education interventions (including e-health platform assistance) for women. Randomized controlled trials (RCT) will be used to test nursing education interventions using a double-blind trial system. (Including e-health platform assistance) Effectiveness, in order to provide simple and fast self-health monitoring and management for the people, and it is expected that the case can early prevent the occurrence of related diseases and ensure the safety of the living environment.

ELIGIBILITY:
Inclusion Criteria:

* (1) Females who are 20 years or older (inclusive); (2) Clear consciousness and no mental disorders; (3) Those who can communicate with others in Mandarin or Taiwanese, are willing to participate in this research after explanation, and sign the consent form.

Exclusion Criteria:

* (1) Diagnosed with mental illness, (2) Cognitive impairment, (3) Under 20 years old, (4) Male.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Basic Demographic Health Assessment Form | baseline, pre-intervention(T0)
  Number, age, gender, marriage, current living area, height, weight, blood pressure, pulse, waist circumference, BMI, education level, past medical history, work-related, living habits, weight control, eating habits; B. Emotional state; C. Female Related questions: menstrual history, fertility status, medication, supplement status, disease history, etc.
.The Environmental Hormone-Plasticizer Health Literacy Scale | baseline, pre-intervention(T0)
  It is divided into three areas of environmental hormone health literacy: Health care, Disease prevention and Health promotion. The answers are based on a Likert 4-point scale, ranging from "very difficult" (1) to "very easy" (4). A higher total score, indicates better environmental hormone-plasticizer health literacy. The total score range is 0-40.
The Environmental Hormone-Plasticizer Health Literacy Scale | three month after intervention(T1)
  It is divided into three areas of environmental hormone health literacy: Health care, Disease prevention and Health promotion. The answers are based on a Likert 4-point scale, ranging from "very difficult" (1) to "very easy" (4). A higher total score, indicates better environmental hormone-plasticizer health literacy. The total score range is 0-40.
The Environmental Hormone-Plasticizer Health Literacy Scale | six month after intervention(T2)
  It is divided into three areas of environmental hormone health literacy: Health care, Disease prevention and Health promotion. The answers are based on a Likert 4-point scale, ranging from "very difficult" (1) to "very easy" (4). A higher total score, indicates better environmental hormone-plasticizer health literacy. The total score range is 0-40.

SECONDARY OUTCOMES:
The System Usability Scale | six month after intervention(T2)] for Experimental arm
  System Usability Scale ( SUS) has ten items, created by John Brooke in 1986 (Brooke, 1986), and is widely used to quickly test standardized questionnaires (objectivity, universality, Repeatable and quantifiable) (Brooke, 2013). Using Likert's five-point scale, questions 1, 3, 5, 7, and 9 are positive questions, and questions 2, 4, 6, 8, and 10 are negative questions. After calculating the scores for each question, multiply all the scores by 2.5 to get the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jung Hsieh, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chuang SC, Chen HC, Sun CW, Chen YA, Wang YH, Chiang CJ, Chen CC, Wang SL, Chen CJ, Hsiung CA. Phthalate exposure and prostate cancer in a population-based nested case-control study. Environ Res. 2020 Feb;181:108902. doi: 10.1016/j.envres.2019.108902. Epub 2019 Nov 8. PMID 31785779
- [Background] Den Hond E, Govarts E, Willems H, Smolders R, Casteleyn L, Kolossa-Gehring M, Schwedler G, Seiwert M, Fiddicke U, Castano A, Esteban M, Angerer J, Koch HM, Schindler BK, Sepai O, Exley K, Bloemen L, Horvat M, Knudsen LE, Joas A, Joas R, Biot P, Aerts D, Koppen G, Katsonouri A, Hadjipanayis A, Krskova A, Maly M, Morck TA, Rudnai P, Kozepesy S, Mulcahy M, Mannion R, Gutleb AC, Fischer ME, Ligocka D, Jakubowski M, Reis MF, Namorado S, Gurzau AE, Lupsa IR, Halzlova K, Jajcaj M, Mazej D, Tratnik JS, Lopez A, Lopez E, Berglund M, Larsson K, Lehmann A, Crettaz P, Schoeters G. First steps toward harmonized human biomonitoring in Europe: demonstration project to perform human biomonitoring on a European scale. Environ Health Perspect. 2015 Mar;123(3):255-63. doi: 10.1289/ehp.1408616. Epub 2014 Dec 11. PMID 25493439
- [Background] Fisher JS. Environmental anti-androgens and male reproductive health: focus on phthalates and testicular dysgenesis syndrome. Reproduction. 2004 Mar;127(3):305-15. doi: 10.1530/rep.1.00025. PMID 15016950
- [Background] Fu Z, Zhao F, Chen K, Xu J, Li P, Xia D, Wu Y. Association between urinary phthalate metabolites and risk of breast cancer and uterine leiomyoma. Reprod Toxicol. 2017 Dec;74:134-142. doi: 10.1016/j.reprotox.2017.09.009. Epub 2017 Sep 23. PMID 28951174
- [Background] Jacobs RJ, Lou JQ, Ownby RL, Caballero J. A systematic review of eHealth interventions to improve health literacy. Health Informatics J. 2016 Jun;22(2):81-98. doi: 10.1177/1460458214534092. Epub 2014 Jun 10. PMID 24916567
- [Background] Wang IJ, Karmaus WJ, Chen SL, Holloway JW, Ewart S. Effects of phthalate exposure on asthma may be mediated through alterations in DNA methylation. Clin Epigenetics. 2015 Mar 15;7(1):27. doi: 10.1186/s13148-015-0060-x. eCollection 2015. PMID 25960783
- [Background] Williams MJ, Wiemerslage L, Gohel P, Kheder S, Kothegala LV, Schioth HB. Dibutyl Phthalate Exposure Disrupts Evolutionarily Conserved Insulin and Glucagon-Like Signaling in Drosophila Males. Endocrinology. 2016 Jun;157(6):2309-21. doi: 10.1210/en.2015-2006. Epub 2016 Apr 21. PMID 27100621
- [Background] Benjamin S, Masai E, Kamimura N, Takahashi K, Anderson RC, Faisal PA. Phthalates impact human health: Epidemiological evidences and plausible mechanism of action. J Hazard Mater. 2017 Oct 15;340:360-383. doi: 10.1016/j.jhazmat.2017.06.036. Epub 2017 Jun 19. PMID 28800814
- [Background] Sharma S, Ashley JM, Hodgson A, Nisker J. Views of pregnant women and clinicians regarding discussion of exposure to phthalate plasticizers. Reprod Health. 2014 Jun 21;11:47. doi: 10.1186/1742-4755-11-47. PMID 24952638